CLINICAL TRIAL: NCT01640990
Title: A Single-centre, Escalating Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Slow Intravenous Infusion of GW328267X in Healthy Volunteers
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of an Intravenous Infusion of GW328267X in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 115387
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Lung Injury, Acute
Keywords: Healthy male volunteers, intravenous infusion, GW328267X, dose escalation,
MeSH Terms: conditions — Acute Lung Injury | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): slow IV infusion over 6 hours consisting of saline for 30 minutes (run in period), 8 mcg/h GW328267X for 1.5 hours (total dose of 12mcg), and 10 mcg/h GW328267X for 4 hours (total dose of 40 mcg)
  Interventions: Drug: Saline; Drug: GW328267X (total dose of 12mcg); Drug: GW328267X (total dose of 40mcg)
- Cohort 2 (Experimental): Dose to be determined after analysis of Cohort 1
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — 30mins run-in period
Drug: GW328267X (total dose of 12mcg) — 8 mcg/h for 1.5 hours (total dose of 12mcg)
  Arms: Cohort 1
Drug: GW328267X (total dose of 40mcg) — 10 mcg/h for 4 hours (total dose of 40 mcg)
  Arms: Cohort 1

SUMMARY:
This study is a single dose evaluation using an open label dose escalating design. Cohort1 will consist of 3 healthy male volunteers. Each volunteer will receive a slow IV infusion over 6 hours consisting of saline for 30 minutes (run in period), 8 mcg/h GW328267X for 1.5 hours (total dose of 12mcg) and 10 mcg/h GW328267X for 4 hours (total dose of 40 mcg). Subjects will have continuous cardiac monitoring throughout the dosing period and up to 2 hours after cessation of the intravenous infusion. PK measurements and measurement of erythropoietin and platelet activation will also be done. Samples for PK will be taken at 30 minute intervals during the infusion of GW328267X up to and including 1 hour after cessation of the intravenous infusion. Samples for erythropoietin and platelet aggregation will be done.

Cohort 2 is optional and may be carried out in the event that the dose of GW328267X given in Cohort 1 is both well tolerated and subjects do not meet the stopping criteria. The decision to proceed to Cohort 2 and the dose level will be made by the GSK Study Team and the Investigator based on safety, tolerability and preliminary PK/PD data obtained in Cohort 1. It is planned that the maximum total dose given to any subject will not exceed 150mcg. Cohort 2 will consist of 3 healthy male volunteers and the study procedures for this additional Cohort will be the same as that described for Cohort 1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male, between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Body weight ≥ 50 kg and BMI within the range 18.5 - 29.9 kg/m2 (inclusive).
* Heart rate within the range 50 - 85 bpm (inclusive) and blood pressure range between 115/60 - 140/90 mmHg (inclusive) at Screening and Day 1.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Single QTcF < 450 msec.
* 24-hour Holter monitoring at screening within normal limits.
* Peripheral veins suitable for venous blood sampling and cannulation

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Have history of any pre-existing cardiac arrhythmias (including sinus tachycardia, atrial fibrillation or flutter) or finding on baseline examination that, in the opinion of the investigator, may place the subject at an unacceptable risk as a participant in this trial or may interfere with interpretation of cardiovascular safety results during the conduct of the trial.
* Current or history of asthma (with the exception of a history of asthma in childhood only).
* Urinary cotinine levels indicative of smoking or a history of regular use of tobacco nicotine-containing products within 6 months prior to screening.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, with the exception of simple analgesics but including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-11-22 (Actual); Primary Completion 2011-12-09 (Actual); Study Completion 2011-12-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability including number of subjects with adverse events assessment | baseline, Day 1, Day 2 and Day 10
Safety and tolerability including change from baseline and number subjects with abnormal clinical safety laboratory data | baseline, Day 1, Day 2 and Day 10
Safety and tolerability, including change from baseline and number of subjects with abnormal ECG assessments | baseline, Day 1, Day 2 and Day 10
Safety and tolerability, including change from baseline and number of subjects with abnormal vital signs (blood pressure and heart rate) assessments | baseline, Day 1, Day 2 and Day 10

SECONDARY OUTCOMES:
Heart rate changes from baseline during intravenous infusion of GW328267X | baseline, Day 1, Day 2 and Day 10
Platelet aggregation parameters | Pre-dose, Day 1 5.5 hr, Day 2
Erythropoietin levels | Screening, Pre-dose, Day 2, Follow Up
Levels of GW328267X in plasma | baseline, Day 1 and Day 2 (24hrs)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115387 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115387?search=study&study_ids=115387#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 115387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115387 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register